CLINICAL TRIAL: NCT00723307
Title: A Randomised Placebo-controlled Trial of Metformin on Progression of Carotid Atherosclerosis in Non-diabetic Patients With Cardiovascular Disease Treated With Conventional Risk Reducing Agents
Brief Title: Carotid Atherosclerosis: MEtformin for Insulin ResistAnce Study
Acronym: CAMERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Naveed Sattar (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor-Investigator, Professor Naveed Sattar, Professor of Metabolic Medicine, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gla-Met-1 (version 5)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: No diabetes mellitus; Elevated waist circumference
MeSH Terms: conditions — Coronary Artery Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — White film-coated tablets, 850mg tablet twice daily, 1.5 years duration
  Other Names: Glucophage; Glucophage SR; Bolamyn SR
  Arms: Metformin
Drug: Placebo — White coated tablet; one tablet twice daily; 1.5 years duration
  Other Names: Dummy pill
  Arms: Placebo

SUMMARY:
Hypothesis: Treatment with metformin in overweight non-diabetic individuals with coronary heart disease and on standard cardiovascular risk reducing agents including statins will have a beneficial impact on carotid artery atherosclerosis compared to placebo.

Rationale: Once subjects have a heart attack, they remain at much higher than average risk of another heart attack and stroke, despite the best current therapies to lower their cholesterol and blood pressure and thin their blood. Many subjects with heart disease also have problems metabolising (i.e. processing) sugar even if they do not have diabetes. There is some evidence that metformin, a drug which improves sugar metabolism, decreases the risk of future heart attacks in diabetic patients. However, whether metformin further reduces the risk of heart disease beyond established treatments in people without diabetes is unknown.

Method: The investigators will test the ability metformin, a drug with proven safety, to slow the progression of furring up (known as atherosclerosis) of blood vessels in non-diabetic subjects with heart disease. This will be achieved by treating 2 groups of subjects with metformin and placebo pills respectively. To measure atherosclerosis, the investigators will carry out ultrasound scans of the big blood vessels in the neck at the start of the study, after 1 year and after 1.5 years of therapy.The investigators will then be able to assess whether metformin has had a beneficial impact.

ELIGIBILITY:
Inclusion Criteria:

* Proven coronary heart disease (prior acute coronary syndrome, prior CABG or angiographically proven CHD)
* Aged 35-75 years
* Elevated waist circumference as per the International Diabetes Foundation criteria (94 cm in men and 80 cm in women)
* All patients will be on statin

Exclusion Criteria:

* Pregnancy and/or lactation at screening
* Premenopausal woman not on contraception
* Known or newly diagnosed diabetes mellitus on oral glucose tolerance testing (OGTT will be performed on subjects with HbA1C 6.0-6.9% and fasting plasma glucose [FPG] < 7.0 mmol/L at screening18)
* Screening results: HbA1C ≥ 7.0% and/or fasting plasma glucose ≥ 7.0 mmol/L
* Patients with Acute Coronary Syndrome within the last 3 months
* Clinically unstable heart failure
* Uncontrolled angina
* Contraindications to metformin

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in progression of carotid intima-media thickness (measured in millimetres) between groups treated with metformin and placebo | 1.5 years

SECONDARY OUTCOMES:
Correlation of HbA1C, t-PA, CRP, IL-6, HOMA-IR and ICAM-1 with change in carotid IMT in metformin- and placebo-treated groups will be evaluated. | 1.5 years
Difference in progression of carotid total plaque area (measured in square millimetres) between groups treated with metformin and placebo | 1.5 years
Difference in progression of carotid total plaque volume (measured in cubic millimetres) between groups treated with metformin and placebo | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Glasgow Clinical Research Facility, NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

REFERENCES:
- [Derived] Preiss D, Welsh P, Sattar N. Metformin Therapy and Circulating NT-proBNP Levels: The CAMERA Trial. Diabetes Care. 2016 Aug;39(8):e114-5. doi: 10.2337/dc16-0887. Epub 2016 Jun 6. No abstract available. PMID 27271181
- [Derived] Preiss D, Lloyd SM, Ford I, McMurray JJ, Holman RR, Welsh P, Fisher M, Packard CJ, Sattar N. Metformin for non-diabetic patients with coronary heart disease (the CAMERA study): a randomised controlled trial. Lancet Diabetes Endocrinol. 2014 Feb;2(2):116-24. doi: 10.1016/S2213-8587(13)70152-9. Epub 2013 Nov 7. PMID 24622715